CLINICAL TRIAL: NCT00980408
Title: The NMDA Receptor Co-agonist D-cycloserine Accelerates Associative Learning in the Human Hippocampal CA Region
Brief Title: The Influence of Glutamate on Memory in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, MD, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RH999
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Individuals
MeSH Terms: interventions — Sugars; Cycloserine; Glutamic Acid; Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Sugar pill, behavioral glutamic acid (Placebo Comparator): Placebo condition for D-Cycloserine
  Interventions: Drug: Sugar pill
- Sugar pill, fMRI, glutamic acid (Placebo Comparator): Placebo condition for D-Cycloserine, fMRI
  Interventions: Drug: Sugar pill
- Sugar pill, memantine, behavioral (Placebo Comparator): Placebo condition Memantine, behavioral
  Interventions: Drug: Sugar pill
- Sugar pill, memantine, fMRI (Placebo Comparator): Placebo condition Memantine, fMRI
  Interventions: Drug: Sugar pill
- D-Cycloserine behavioral (Active Comparator)
  Interventions: Drug: Glutamic Acid
- D-Cycloserine, fMRI (Active Comparator)
  Interventions: Drug: Glutamic Acid
- Memantine, behavioral (Active Comparator)
  Interventions: Drug: Memantine
- Memantine, fMRI (Active Comparator)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Sugar pill — 250 mg, one dose, 60 min prior
  Other Names: Placebo condition for D-Cycloserine, behavioral study
  Arms: Sugar pill, behavioral glutamic acid
Drug: Sugar pill — 250 mg, one dose, 60 min prior
  Other Names: Placebo condition for D-Cycloserine, fMRI
  Arms: Sugar pill, fMRI, glutamic acid
Drug: Sugar pill — 20 mg, one dose, 8 hours prior
  Other Names: Placebo condition Memantine, behavioral
  Arms: Sugar pill, memantine, behavioral
Drug: Sugar pill — 20 mg, one dose, 8 hours prior
  Other Names: Placebo condition Memantine, fMRI
  Arms: Sugar pill, memantine, fMRI
Drug: Glutamic Acid — 250 mg, one dose, 60 minutes prior
  Other Names: D-Cycloserine, King Pharmaceuticals
  Arms: D-Cycloserine behavioral
Drug: Glutamic Acid — 250 mg, one dose, 60 minutes prior
  Other Names: D-Cycloserine, King Pharmaceuticals
  Arms: D-Cycloserine, fMRI
Drug: Memantine — 20 mg, one dose, 8 hours prior
  Other Names: Axura, Merz
  Arms: Memantine, behavioral
Drug: Memantine — 20 mg, one dose, 8 hours prior
  Other Names: Axura, Merz
  Arms: Memantine, fMRI

SUMMARY:
The hippocampus is particularly laden with n-methyl-d-aspartate (NMDA) receptors, and is at the same time one of the most important sites in declarative memory. The rationale of this study is that the NMDA partial agonist D-Cycloserine will promote learning compared to a placebo. On the other hand, the NMDA receptor antagonist Memantine might lead to reduced memory. We believe that the influence of NMDA receptors on memory can be determined via acute co-activation of the NMDA receptors with Cycloserine® (King Pharmaceuticals Ltd, active ingredient: DCycloserin, dose: 250 mg) and Memantine (Axura®, Merz, active ingredient: Memantine, dose: 20 mg)on both a behavioral and functional (fMRI) level.

ELIGIBILITY:
Inclusion Criteria:

* German native language or native language level
* Able to give written informed consent
* right-handed

Exclusion Criteria:

* inability to give written informed consent, underaged minors, contractually incapable persons, persons in legal custody
* any psychiatric, neurological or internal illness
* hematoporphyria (enzyme sickness)
* intake of medication (except oral contraceptives)
* simultaneous participation in other clinical studies
* hypersensitivity to Memantine or other anti-dementia substances, or to D-Cycloserine
* alcohol abuse
* epilepsy
* depression
* serious anxiety or psychosis
* serious kidney insufficiency
* intake of Ethionamide or Isoniazide
* pregnancy or women who are nursing
* liver or kidney problems
* intake of NMDA-antagonists, such as Amantadine, Ketamine, or Dextromethorphan
* vegetarians
* stomach ulcer, if treated with medication
* renal tubular acidosis
* urinary infections (with proteus bacteria)
* recent heart attack, heart failure, or uncontrolled high blood pressure
* intake of L-Dopa, dopaminergic agonists, and anticholinergics
* intake of barbiturates, spasmolytics, Phenytoin, Amantadine, oral coagulators, warfarin, HCT (Hydrochlorothiazide)
* heart or cranial operations
* pacemaker, medication pump (such as insulin pump), hearing aid, removable prosthodontics
* metal in or on body (such as acupuncture needles, artificial limbs, stents, metal splints, clips, implanted electrodes, tattoos, or piercings)
* claustrophobia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
fMRI during learning task | once at drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Forschungszentrum Juelich GmbH, Jülich, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Onur OA, Schlaepfer TE, Kukolja J, Bauer A, Jeung H, Patin A, Otte DM, Shah NJ, Maier W, Kendrick KM, Fink GR, Hurlemann R. The N-methyl-D-aspartate receptor co-agonist D-cycloserine facilitates declarative learning and hippocampal activity in humans. Biol Psychiatry. 2010 Jun 15;67(12):1205-11. doi: 10.1016/j.biopsych.2010.01.022. Epub 2010 Mar 20. PMID 20303474